CLINICAL TRIAL: NCT07385222
Title: A Single-Center Prospective Interventional Study Comparing Pelvic Floor Muscle Training Alone Versus Combined With Extracorporeal Magnetic Innervation in Men With Premature Ejaculation
Brief Title: Pelvic Floor Muscle Training With or Without Extracorporeal Magnetic Innervation for Premature Ejaculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Fatih UYSAL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-MFU-01
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-01

CONDITIONS: Premature (Early) Ejaculation; Ejaculatory Dysfunction; Sexual Dysfunction Male
Keywords: premature ejaculation; pelvic floor; pelvic floor muscle training; magnetic field therapy; ultrasonography
MeSH Terms: conditions — Premature Birth; Ejaculatory Dysfunction; Premature Ejaculation

STUDY DESIGN:
Intervention Model Description: parallel-group controlled interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Pelvic Floor Muscle Training (PFMT) (Active Comparator): Structured pelvic floor education plus a progressive home exercise program supervised during the 8-week period.
  Interventions: Behavioral: Pelvic Floor Muscle Training
- Arm B - Pelvic Floor Muscle Training (PFMT) + Extracorporeal Magnetic Innervation (ExMI) (Experimental): PFMT as in Arm A, plus chair-based magnetic stimulation delivered per predefined clinic protocol over 8 weeks.
  Interventions: Behavioral: Pelvic Floor Muscle Training; Device: Extracorporeal Magnetic Innervation

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training — Structured pelvic floor education plus a progressive home exercise program supervised during the 8-week period.
Device: Extracorporeal Magnetic Innervation — PFMT as in Arm A, plus chair-based magnetic stimulation delivered per predefined clinic protocol over 8 weeks.
  Arms: Arm B - Pelvic Floor Muscle Training (PFMT) + Extracorporeal Magnetic Innervation (ExMI)

SUMMARY:
This is a single-center, prospective interventional study comparing pelvic floor muscle training (PFMT) alone versus PFMT combined with extracorporeal magnetic innervation (ExMI) in men with premature ejaculation (PE). The objective was to determine whether adding ExMI to standard PFMT improves pelvic floor function and patient-reported sexual outcomes.

DETAILED DESCRIPTION:
This is a single-center, prospective interventional study that prospectively evaluated two nonpharmacological approaches for the management of premature ejaculation (PE): pelvic floor muscle training (PFMT) alone versus PFMT combined with extracorporeal magnetic innervation (ExMI). Adult men with clinically diagnosed PE were enrolled at a university hospital physiotherapy/urology clinic and followed over an 8-week intervention period. The trial was open-label with parallel groups; participants received the treatment used in clinical practice (PFMT only or PFMT+ExMI), and outcomes were collected prospectively according to a predefined protocol.

PE is common and impairs quality of life. PFMT may improve neuromuscular control of the pelvic floor, and ExMI delivers chair-based magnetic stimulation to activate pelvic floor musculature. We hypothesized that adding ExMI to standard PFMT would produce greater improvements in pelvic floor function and patient-reported sexual outcomes than PFMT alone.

All participants received structured education and a progressive, home-based PFMT program supervised during the 8-week period. The PFMT+ExMI group additionally underwent chair-based magnetic stimulation delivered per the clinic's predefined protocol targeting pelvic floor muscles.

Assessments were performed at baseline and post-intervention (week 8), with short-term follow-up where feasible. Primary outcomes were pelvic floor muscle displacement distance and endurance measured with real-time suprapubic ultrasonography under standardized instructions. Secondary outcomes included the Premature Ejaculation Diagnostic Tool (PEDT), International Index of Erectile Function (IIEF-5), Male Sexual Function Inventory-Short Form (MSFI-SF), WHOQOL-BREF sexual satisfaction item, Global Perceived Effect, and safety/adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male, 25-45 years, sexually active
* Clinical diagnosis of premature ejaculation by a specialist
* Able to comply with PFMT and assessments
* Complete baseline clinical/ultrasound records

Exclusion Criteria:

* Neurologic disease (e.g., multiple sclerosis)
* Metabolic/systemic/psychiatric disorders impacting outcomes
* Significant cardiovascular disease
* Medications affecting erection/ejaculation
* Chronic prostatitis/urethritis or active UTI
* Peyronie's disease or prior penile prosthesis at baseline

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male only.
Enrollment: 41 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle displacement distance (mm) on real-time suprapubic ultrasonography | Baseline, Week 4 and Week 8 (post-intervention)
  Change from baseline in cranio-caudal displacement during standardized contraction.
Pelvic floor muscle endurance (seconds) on real-time suprapubic ultrasonography | Baseline, Week 4 and Week 8
  Change from baseline in sustained contraction time under standardized instruction.

SECONDARY OUTCOMES:
Premature Ejaculation Diagnostic Tool | Baseline, Week 4 and Week 8
  This five-item, Likert-type self-report form measures the severity of premature ejaculation by assessing ejaculation control, intravaginal ejaculation time, and emotional impact.
Male Sexual Function Inventory-Short Form | Baseline, Week 4 and Week 8
  This instrument evaluates male sexuality in terms of functional domains and allows for the analysis of psychometric properties related to overall sexual satisfaction. Each item is rated on a Likert scale ranging from 0 (dysfunction/severe problem) to 4 (good function/no problem)
International Index of Erectile Function | Baseline, Week 4 and Week 8
  This self-assessment tool is widely used to determine the severity of erectile dysfunction.
World Health Organization Quality-of-Life Scale-BREF | Baseline, Week 4 and Week 8
  This tool enables individuals to subjectively assess their quality of life in physical, psychological, social, and environmental domains within their own cultural context.
Global Perceived Effect Scale | at Week 8
  This scale aims to measure how individuals experience recovery processes in relation to factors such as health status, emotional state, perceived stress, and social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No